CLINICAL TRIAL: NCT03630523
Title: Registering the Immune Response to a Flu Vaccination Challenge in PTEN Hamartoma Tumour Syndrome
Brief Title: Response of Immune System to Flu Vaccination in PHTS
Acronym: RIPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL66559.091.18
Record Dates: First submitted 2018-08-10; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: PTEN Hamartoma Tumor Syndrome
Keywords: PHTS; PTEN; Vaccination
MeSH Terms: conditions — Hamartoma Syndrome, Multiple

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccination (Other): Arm contains all subjects; vaccination with Influvac Tetra will be administered at start of study, response will be measured in 7 and 21 days.
  Interventions: Biological: Influvac Tetra

INTERVENTIONS:
Biological: Influvac Tetra — Tetravalent seasonal flu vaccination 2018/2019

SUMMARY:
this study evaluates the cellular and humoral immune response to seasonal influenze vaccination in PTEN Hamartoma Tumor Syndrome. All subjects will be administered flu vaccination, half of the subjects will be control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with PHTS based on genetic testing
* Must be a Radboudumc patient
* Must be 18 years or older
* Must be mentally competent
* Must have provided written informed consent to participate in the study
* Must be able to adhere to visit schedule and available to complete the study

Exclusion Criteria:

* • Known history of significant medical disorder, which in the investigator's judgment might confound the results of the study or pose additional risk to the subject by participation in the study

  * Known hypersensitivity to previous influenza vaccinations (Anaphylaxis)
  * Must not be allergic to chicken eggwhite
  * Pregnancy at start of study
  * Immunocompromised patients and those receiving concomitant immunosuppressive therapy or other immune modulating drugs including chronic steroid treatment.
  * Bleeding disorders including haemophilia and thrombocytopenia or treatment with anticoagulants(Due to risk of intramuscular hematoma after injection)
  * Must not have received vaccination with attenuated pathogens in the 4 weeks leading up to study. (Measles, mumps, rubella, yellow fever, rotavirus, BCG, typhoid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Hemagglutination inhibition assay titre | 7 days

SECONDARY OUTCOMES:
Proliferation assay | 21 days
interleukin profile | 21 days, 7 days